CLINICAL TRIAL: NCT00775918
Title: Single Dose Two-Way Crossover Fed Bioequivalence Study of Doxycycline Monohydrate 100 mg Tablets in Healthy Volunteers
Brief Title: Bioequivaelnce Study of Doxycycline Monohydrate 100mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Laboratories Limited
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AAI-US-312
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence Doxycycline monohydrate 100mg tablets fed conditions
MeSH Terms: interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Doxycycline monohydrate 100mg tablets of Ranbaxy
  Interventions: Drug: Doxycycline monohydrate 100mg tablets
- 2 (Active Comparator): Adoxa ® 100 mg tablets of Bradley Pharmaceuticals Inc
  Interventions: Drug: Doxycycline monohydrate 100mg tablets

INTERVENTIONS:
Drug: Doxycycline monohydrate 100mg tablets — Bioequiavelnce Doxycycline monohydrate 100mg tablets fed conditions

SUMMARY:
The purpose of this study was to determine the bioequivalence of Doxycycline monohydrate formulations after administration of single doses to normal healthy subjects under fed conditions. These data were to be evaluated statistically to determine if the products meet bioequivalence criteria.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomised, two-treatment, two-period, two-sequence, single-dose, crossover , bioequivalence study on Doxycycline monohydrate comparing Doxycycline monohydrate 100mg tablets of Ranbaxy Pharmaceuticals Inc with Adoxa ® 100 mg tablets of Bradley Pharmaceuticals Inc. in healthy, adult, human, subjects under fed conditions.

A total of 32 non-smoking subjects (21 men and 11 women) were included in this study, of which 32 finished the study according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* a) Healthy male and female subjects of at least 18 years of age. b) Informed of the nature of the study and given written informed consent. c). Have a body mass index between 18 and 30 and weighing at least 110 pounds. d) In good health as determined by lacking of clinically significant abnormalities in health assessments performed at screening as judged by the physician.

Exclusion Criteria:

* a) Hypersensitivity to Doxycycline monohydrate (Adoxa®), or related compounds such as tetracycline.

  b) Any history of a clinical condition which might affect drug absorption, metabolism or passage of drugs out of the body, e.g. sprue, celiac disease, Crohn's disease, colitis, liver, kidney or thyroid conditions.

  c) Recent history of mental illness, drug addiction, drug abuse or alcoholism. d) Donation of greater than 500 ml of blood in the past 4 weeks prior to study dosing or difficulty in donating blood.

  e) Received an investigational drug within the 4 weeks prior to study dosing. f) Currently taking any systemic prescription medication, except oral / cutaneous/ vaginal hormone contraceptives, within the 7 days prior to study dosing or over-the-counter medication within 3 days of study dosing. This prohibition does not include vitamins or herbal preparations taken as nutritional supplements for non-therapeutic indications as judged by the attending physician. Any non-prescription medication consumption reported will be reviewed by the investigator prior to dosing. At the discretion of the investigator these volunteers may be enrolled if the medication is not anticipated to alter study integrity.

  g) Regular smoking of more than 5 cigarettes per week or the daily use of nicotine-containing products beginning 3 months before the study medication administration through the final evaluation.

  h) If female, the subject is lactating or has a positive pregnancy test at screening and prior to each of the two treatment periods. Females of child bearing potential must use a 'medically acceptable method of contraception throughout the entire study period and for one week after the study is completed. Medically acceptable methods of contraception that may be used by the subject and/or her partner are: oral contraceptives/ patches, progestin injection or implants, condom with spermicide, diaphragm with spermicide, IUD, vaginal spermicidal or hormonal suppository, surgical Sterilization of themselves or their partner(s) or abstinence. Females taking oral Contraceptives must have taken them consistently for at least three months prior to receiving study medication.

  i) Alcohol, grapefruit beverages or foods or caffeine beverages or foods beginning 24 hours before each study medication administration through each study confinement period. Such restricted items include tea, coffee, iced tea, coke, Pepsi, mountain dew, chocolate, brownies, etc.

  j) Significant history or current evidence of chronic infectious disease, system disorders or organ dysfunction k) Regular use of any drugs known to induce or inhibit hepatic drug metabolism (e.g. barbiturates, carbamazepine, rifampin, phenylhydantaoins, phenothiazines, cimetidine, Omeprazole, macrolides, imidazoles, fluoroquinolines) within 30 days prior to study administration l) Positive test results for HIV, hepatitis B surface antigen, hepatitis C antibodies, drugs of abuse, or pregnancy at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-06; Primary Completion 2005-06 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- aaiPharma, Inc., Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html